CLINICAL TRIAL: NCT07136753
Title: The IMpact of 3D Surface Imaging and Simulation on Shared Decision Making in Immediate Breast REconstruction And the Measurement of the EffectS of RadioTherapy
Brief Title: MIBREAST Making in Immediate Breast REconstruction And the Measurement of the EffectS of RadioTherapy
Acronym: MIBREAST
Status: Recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5635
Record Dates: First submitted 2025-02-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Decision making; Reconstruction; Risk reducing surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of Care: 2D catalogue of photographs of other patients who have had surgery to demonstrate the predicted post-operative appearance
- 3D Surface Imaging: 3D Simulation of patients own breast to show them how they might look after surgery

SUMMARY:
Patients who require a removal of a breast (mastectomy) for breast cancer or future risk reduction often have immediate breast reconstruction (IBR). This can be performed using either an implant or the patient's own body fat to recreate the breast shape.

Patients can find it difficult to imagine their own post-surgery appearance. Using 3D surface imaging (3D-SI) can change a patient's pictures to show them how they might look after surgery, known as a simulation. Some patients may find 3D-SI and simulation gives them confidence in their expectations and others may not feel it helps much.

This study will investigate the following 3 questions:

1. Whether 3D-SI and simulation can improve patient confidence about their likely post-surgery appearance
2. Whether 3D-SI measurement of breast shape helps in surgical planning and reduces the need for later adjustment surgery to improve symmetry, especially in patients having a mastectomy on one side only
3. How much radiotherapy changes breast reconstructions over time using 3D- SI to objectively measure this. For this study the follow up for some women who do and some who do not have radiotherapy after breast reconstruction.

3D surface imaging may improve surgeon understanding of breast shape, prior to surgery. In cases where there is a high risk of breast cancer recurrence patients are offered radiotherapy to the breast, either before or after surgery. Radiotherapy has a negative impact on the reconstructed breast, and may cause it to shrink and change position but the effect of radiotherapy has never been accurately quantified. This study will be investigating the following:

1. Whether 3D-SI measurement of breast shape helps in surgical planning and reduces the need for later adjustment surgery to improve symmetry, especially in patients having a mastectomy on one side only
2. How much radiotherapy changes breast reconstructions over time using 3D- SI to objectively measure this. For this study the follow up some women who do and some who do not have radiotherapy after breast reconstruction.

DETAILED DESCRIPTION:
Approximately 40% of all women diagnosed with breast cancer (BC) will require a mastectomy and a large proportion (60%) of these will choose to have an immediate breast reconstruction (IBR).

Patient satisfaction with physical appearance after completion of their BC treatment has a well-documented association not only with their psychological wellbeing but also improved quality of life. Due to advances in oncological therapies, BC patients now have excellent survival rates of 85% at five years and 75% at ten years meaning that more women survive to experience the long-term impact of surgical and radiotherapy treatments and highlights the importance of improving aesthetic outcome as a survivorship focus.

3D-surface imaging (3D-SI) and simulation is frequently used to demonstrate cosmetic breast augmentation outcomes in the private sector and is increasingly being used in breast cancer surgery.

Effective communication of the post-operative aesthetic outcome and the possible requirement of adjustment surgery to patients is a central part of the informed consent process. Women sometimes struggle to decide between breast-conserving treatment and mastectomy with or without reconstruction. Those that want reconstruction to have the option of using a silicone implant, or their own tissue, transplanted from the abdomen or inner thigh (an autologous flap). Consultations focus on the patient's desires and expectations, and the surgeon's explanation of what is technically possible, the benefits and compromises, until a mutual understanding is reached. This can however be challenging, particularly when attempting to predict the effects of adjuvant radiotherapy on the reconstructed breast. Traditionally, surgeons have used diagrams or 2D clinical photographs of other patients who have had surgery to demonstrate the predicted post-operative appearance. Many patients have reported that they find these methods unhelpful and confusing, as the wide variety of body habitus, breast shape, skin tone and surgical options mean that it is unlikely that a woman will see images adequately illustrating her own unique outcome.

The hypothesise that viewing 3D simulations of their own likely appearance after mastectomy and breast reconstruction will give women more confidence and certainty as they approach surgery. There are not yet in a position to use 3D-SI as a decision-support tool.

The overarching aim of this study is to evaluate the utility of 3D-SI in simulation and measurement of outcome of immediate breast reconstruction.

Hypothesis 1 - Impact of 3D Simulation on Shared Decision Making Women who see a simulation of their IBR outcome will have more confidence in their decision-making about IBR options.

Hypothesis 2 - Impact of 3D-SI on Elective Surgical Revision rate A better understanding of breast shape may reduce the need for elective surgical revisions such as volume-adjustment procedures (lipofilling or liposuction) in the reconstructed breast.

Hypothesis 3 - Impact of Radiotherapy on IBR The hypothesise that immediate breast reconstructions that receive radiotherapy undergo greater change in shape and position over time.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged > 18
* Undergoing immediate breast reconstruction (autologous or implant based) follow mastectomy for breast cancer or as a risk-reducing strategy
* Available to attend 3D-SI appointments at specified intervals

Exclusion Criteria:

* Lack of capacity
* Language barrier that prevents patients from understanding the English questionnaires
* Visual impairment
* Unable to answer study questionnaires
* Disability that may prevent appropriate positioning during the imaging process
* Unable to attend for photography
* Requiring delayed reconstruction or no longer considering a reconstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only
Study Population: Patients considering breast reconstruction following mastectomy for cancer or risk reduction.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Difference in Visual Analogue Scale Score | Preioperative/Periprocedural
  Difference in mean visual analogue scale (VAS) for the question 'How confident is one in knowing how their breasts are likely to look after treatment?' VAS score is on a scale from 0-10 (0 indicates not at all confident and 10 indicates very confident)

SECONDARY OUTCOMES:
Difference in decisional conflict scale score | Perioperative/Periprocedural
  Difference in Decisional Conflict Scale (DCS) score for women who see and do not see their simulated reconstruction
Comparison between 3D and SoC anthropometric measurements | Perioperative/Periprocedural
  Comparison between Crisalix and routine tape measure anthropometric measurements.The same unit of measurement will be used for the anthropometric distances (i.e.sternal notch to nippple, nipple to nipple, nipple to midline, nipple to lateral fold, nipple to inframammary fold and breast diameter) measured in cm for both 3D-SI and tape measurements
Thematic analysis of surgeons' experience | 1 year
  Thematic analysis of surgeons' experience
Evaluation of actual outcome against simulated appearance by panel assessment using a Likert scale | through study completion, an average of 1 year
  Evaluation of the actual outcome against the simulated appearance
Comparison of patient satisfaction with the breast, and with information given (BREAST-Q domains) by randomisation group | through study completion, an average of 1 year
  Comparison of patient satisfaction with the breast, and with information given (BREAST-Q domains) by randomisation group (3D simulation vs standard of care) at 1 and 2 years. To further undertake a panel assessment of 3D simulated outcomes and compare these to 2D images of actual post-operative appearance at 1 year after surgery. The panel will consist of consultant breast and plastic surgeons who will indicate likeness of simulated appearance to actual appearance on a Likert scale of 1-5 (score of 1 indicates that simulation is not at a similar to actual outcome and 5 indicates very similar appearance).
Using 3D-SI to classify breast shape | through study completion, an average of 1 year
  Using 3D-SI to classify breast shape
Impact of breast shape classification on elective secondary revisions (ESRs) and reconstructive outcomes | through study completion, an average of 1 year
  Impact of breast shape classification on elective secondary revisions (ESRs) and reconstructive outcomes. 3D-SI measurements (distances in cm and volume in cc) will be captured and using a principal component analysis different breast shape subgroups will be derived. Following this, to then compare breast shape type, primary surgery type (e.g. implant or autologous reconstruction) and whether the patient has had elective surgical revision. This will be an exploratory process to determine whether there is a relationship between breast shape and need for revision surgery. There is currently no existing tool to measure this. anthropometric measurements (sternal notch to nipple, nipple to nipple, nipple to inframammary fold, nipple to midline, nipple to lateral fold, breast diameter) are entered in cm and breast volume is entered in cc.
Documented relationship between donor tissue availability and breast volume | through study completion, an average of 1 year
  The intend to examine the relationship between the available abdominal donor tissue and required breast volume for patients undergoing autologous breast reconstruction. A comparison of the available abdominal tissue (measured in cc) using manual segmentation of the CT scan and the required breast volume measured in cc on the pre-operative 3D-SI measurement. We would like to investigate whether a greater degree of mismatch (abdominal volume in cc divided by breast volume in cc) is related to an increased likelihood of requiring revisional surgery.
Documented changes in shape of IBR with and without radiotherapy | through study completion, an average of 1 year
  volume Documented changes in shape of IBR with and without radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No